CLINICAL TRIAL: NCT06516120
Title: Kinematics of Upper Limb Movements Provoked by an Augmented Reality App in Comparison to Therapy Exercises.
Brief Title: Kinematics of Movements Provoked by an Augmented Reality App
Status: Recruiting | Type: Observational
Sponsor: Sint Maartenskliniek (Other)
Collaborators: Eodyne Systems SL (Industry)
Responsible Party: Sponsor
Other Study IDs: 1103
Record Dates: First submitted 2024-03-06; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Healthy Aging
Keywords: Home-based rehabilitation; Augmented reality; Upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy elderly: Group of participants who have no prior history of stroke
  Interventions: Behavioral: RGS-app
- Stroke survivor: Group of participants who have been through a stroke
  Interventions: Behavioral: RGS-app

INTERVENTIONS:
Behavioral: RGS-app — Participants use the RGS-app on a smartwatch once for 1.5 hours during the measurement. The RGS-app consists of augmented reality games to provoke upper limb movement.

SUMMARY:
Introduction: Home-based rehabilitation has the potential to reduce healthcare costs. However, due to less supervision in the home situation, it is possible that movements are made incorrectly. Therefore it is important to gain insight in which movements are made with a home-based rehabilitation system and what effects instructions could have on these movements. The current study investigated these movements made by the Rehabilitation Gaming System (RGS) app, this app uses augmented reality to provoke upper limb movements.

Methods: 16 healthy elderly and 16 stroke survivors participate in this study. Each participant was invited to the rehabilitation clinic for a one time measurement of 1.5 hours. During this measurement, four therapy exercises and four games on the RGS-app are performed. Each game should provoke a similar movement as one of the therapy exercises. Participants start with performing the therapy exercises for two minutes each. Thereafter they receive a video instruction on how to perform one of the games of the RGS-app, and they will play this game for 2 minutes. Thereafter the group is randomized into two conditions. The first group receives the same video instruction, while the second group receives a personalized live instruction based on the first two minutes of playing. After the new instruction, participants will play the game for two minutes again. This is repeated for all four games. Both the order of the therapy exercises and RGS-app games are randomized. During the study, participants wear Inertial Measurement Units (IMU's).

ELIGIBILITY:
Inclusion Criteria stroke survivors:

* People who suffered from a stroke at least 2 months ago.
* Smartphone users
* Mild to moderate upper limb impairment (Medical Research Council Scale for Muscle Strength (MRC) ≥ 2)

Exclusion Criteria stroke survivors:

* Severe cognitive impairment (Montreal Cognitive Assessment < 19)
* Visual impairments (which cannot be corrected with glasses)
* Upper limb impairments not caused by the stroke

Inclusion Criteria healthy elderly:

* 60 years or older
* Smartphone users

Exclusion Criteria healthy elderly:

* Visual impairments (which cannot be corrected with glasses)
* Upper limb impairments which can affect smartphone use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke survivors will be recruited through a Rehabilitation physician at the Sint Maartenskliniek and if needed through social media.
  Healthy elderly will be recruited using social media.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Average movement velocity | Measured when using the RGS-app during the one-time measurement of 1.5 hours
  Average velocity of every 2-minute session. Velocity is measured at the hand relative to the sternum.

SECONDARY OUTCOMES:
Elbow mean angular velocity | Measured when using the RGS-app during the one-time measurement of 1.5 hours
  Mean angular velocity in m/s of the elbow joint
Pelvis mean angular velocity | Measured when using the RGS-app during the one-time measurement of 1.5 hours
  Mean angular velocity will be calculated in m/s of the pelvis joint
Elbow Range of motion | Measured when using the RGS-app during the one-time measurement of 1.5 hours
  Range of motion in degrees of the elbow joint (0 degrees being fully stretched)
Pelvis range of motion | Measured when using the RGS-app during the one-time measurement of 1.5 hours
  Range of motion in degrees of the elbow joint (0 degrees meaning vertical)

CONTACTS AND LOCATIONS:
Overall Officials: Noël Keijsers, Prof., Principal Investigator — Donders Institute for Brain, Cognition and Behavior, Radboud University
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No